CLINICAL TRIAL: NCT03116308
Title: Effect of Food on Opicapone Bioavailability and Pharmacodynamics in Healthy Subjects
Brief Title: Effect of Food on Opicapone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-91067-128
Record Dates: First submitted 2017-04-12; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 50 mg OPC (Experimental): Subjects received 50 mg OPC once-daily in the evening for 12 days. On D9 subjects were to receive 50 mg OPC in the evening after a minimum 6 hours fast. On D10 subjects were to receive the QD dose of 50 mg OPC thirty minutes after the start of moderate meal (with a previous 6 hours fast)
  Interventions: Drug: Opicapone (OPC)

INTERVENTIONS:
Drug: Opicapone (OPC) — 50 mg OPC capsules; oral route
  Other Names: Ongentys; BIA 9-1067

SUMMARY:
The purpose of this study is to investigate the effect of food on the catechol-O-Methyltransferase (COMT) activity after repeated doses of opicapone (OPC, development code BIA 9-1067) in healthy subjects and to characterize the effects of food on the pharmacokinetics (PK) and tolerability of OPC after repeated doses.

DETAILED DESCRIPTION:
Single-centre, open-label, single-arm study in 28 healthy subjects. Subjects received a single-dose of 50 mg OPC once-daily (QD) in the evening for 12 days. On Day 1 (D1), 50 mg OPC was orally administered in the evening (reference hour for all other administrations) after a minimum of 6 hours fast. From D2 to D8 subjects were in ambulatory and received 50 mg OPC once-daily (evening administration after 2 hours fast). On D9, 50 mg OPC was orally administered in the evening after a minimum of 6 hours fast. On D10, 50 mg OPC was orally administered in the evening, thirty minutes after the start of a moderate meal (with a previous 6 hours fast). On D11 and D12 subjects received the last doses of 50 mg OPC (evening administration after 2 hours fast).

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent and to comply with the study restrictions.
* Male or female subjects aged between 18 and 45 years, inclusive.
* Body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Negative tests for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab at screening.
* Clinical laboratory test results clinically acceptable at screening and admission.
* Negative screen for alcohol and drugs of abuse at screening and admission.
* Non-smokers or ex-smokers for at least 3 months.
* If female:
* Not of childbearing potential by reason of surgery or, if of childbearing potential, she uses an effective non-hormonal method of contraception (intrauterine device or intrauterine system; condom or occlusive cap [diaphragm or cervical or vault caps] with spermicidal foam or gel or film or cream or suppository; true abstinence; or vasectomized male partner, provided that he is the sole partner of that subject) for all the duration of the study.
* Negative serum pregnancy test at screening and a negative urine pregnancy test on admission.

Exclusion Criteria:

* Clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Clinically relevant surgical history.
* Clinically relevant abnormality in the coagulation tests.
* Clinically relevant abnormality in the liver function tests.
* History of relevant atopy or drug hypersensitivity, particularly to any COMT inhibitor.
* History of alcoholism or drug abuse.
* Consume more than 14 units of alcohol a week.
* Significant infection or known inflammatory process at screening or admission.
* Acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhoea, heartburn) at the time of screening or admission.
* Used medicines within 2 weeks of admission that may affect the safety or other study assessments, in the investigator's opinion.
* Previously received OPC.
* Used any investigational drug or participated in any clinical trial within 90 days prior to screening.
* Participated in more than 2 clinical trials within the 12 months prior to screening.
* Donated or received any blood or blood products within the 3 months prior to screening.
* Vegetarians, vegans or have medical dietary restrictions.
* Cannot communicate reliably with the investigator.
* Unlikely to co-operate with the requirements of the study.
* If female:
* Pregnant or breast-feeding.
* Of childbearing potential and not used an approved effective contraceptive method or she uses oral contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-11-21 (Actual); Primary Completion 2015-01-28 (Actual); Study Completion 2015-01-28 (Actual)

PRIMARY OUTCOMES:
Maximum observed effect on COMT activity (Emax) - Day 9 (fasted state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacodynamic parameters for opicapone
Time to occurrence of Emax (tEmax) - Day 9 (fasted state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacodynamic parameters for opicapone
Area under the effect-time curve (AUEC) - Day 9 (fasted state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacodynamic parameters for opicapone
Maximum observed effect on COMT activity (Emax) - Day 10 (fed state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacodynamic parameters for opicapone
Time to occurrence of Emax (tEmax) - Day 10 (fed state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacodynamic parameters for opicapone
Area under the effect-time curve (AUEC) - Day 10 (fed state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacodynamic parameters for opicapone

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) - Day 9 (fasted state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacokinetic parameters for opicapone
Time of occurrence of Cmax (tmax) - Day 9 (fasted state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacokinetic parameters for opicapone
Maximum observed plasma concentration (Cmax) - Day 10 (fed state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacokinetic parameters for opicapone
Time of occurrence of Cmax (tmax) - Day 10 (fed state) | Before and ½, 1, 2, 3, 4, 6, 12 and 24 h post-dose
  Pharmacokinetic parameters for opicapone

IPD SHARING:
Plan to Share IPD: Undecided